CLINICAL TRIAL: NCT05034705
Title: A Randomised Controlled Clinical Trial on the Use of a Dental Aerosol Box to Prevent Microbial Transmission During Dental Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Wan Nurazreena Wan Hassan, Associate Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSRG001-2020ST
Record Dates: First submitted 2021-07-23; First posted 2021-09-05 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Calculi
MeSH Terms: conditions — Calculi

STUDY DESIGN:
Intervention Model Description: Control - conventional suction system Interventional - dental aerosol box with modified high volume evacuation suction system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active comparator: Conventional suction system (Active Comparator): This is the conventional method of using the dental high volume suction to contain the aerosol generated during dental procedure. The saliva ejector will also be used.
  Interventions: Device: Conventional suction system
- Experimental: Dental aerosol box with modified high volume evacuation system (Experimental): The dental aerosol box will be equipped with an exit for the high volume suction to be attached to contain the aerosol generated during dental procedure. The saliva ejector will also be used.
  Interventions: Device: Dental aerosol box with modified high volume evacuation system

INTERVENTIONS:
Device: Conventional suction system — This is the conventional method of using the dental high volume suction to contain the aerosol generated during dental procedure. The saliva ejector will also be used.
  Arms: Active comparator: Conventional suction system
Device: Dental aerosol box with modified high volume evacuation system — The dental aerosol box will be equipped with an exit for the high volume suction to be attached to contain the aerosol generated during dental procedure. The saliva ejector will also be used.
  Arms: Experimental: Dental aerosol box with modified high volume evacuation system

SUMMARY:
The study compares the use of a dental aerosol box in preventing microbial transmission during dental procedure. Subjects requiring scaling treatment (BPE 2) will be recruited. Subjects will be allocated either into the control group (conventional suction method) or interventional group (dental aerosol box) Treatment will involve scaling of two quadrants, where data collection of the microbes will be taken. Secondary outcome will involve a self-administered questionnaire on patients acceptance over the scaling procedure either with conventional suction or using the dental aerosol box to contain the aerosol generated during the scaling procedure.

DETAILED DESCRIPTION:
A closed operation room, with the facility to fumigate the room is chosen for all treatment procedures. Patients would be treated with time separations that would be reasonable to prevent microbial detection of the previous patient.

Sample size calculated based on Sadun et al (2020) to compare two groups would require 15 subjects per group for a 90% power and 0.05 significance.

Inclusion criteria: BPE 2 on at least 2 quadrants. Exclusion criteria: Smoker and systemic disease.

Patients will be randomised using randomiser.org. The list will be placed in a sealed envelop by an individual not involved in subject recruitment. Patient grouping will be determined after recruitment and consent. The envelop will be opened and patient allocated to the group.

Interventional group:

1. Conventional suction (control)
2. Dental aerosol box with modified high-volume evacuation system (interventional)

The procedure will involve scaling of two quadrants, where data collection of the microbes will be taken.

Before each appointment, at the start of study all operatory surfaces were cleaned and disinfected with Ethyl alcohol (70%). Between each treatment and at start of treatment, ultrasonic scaler units will be flushed with water for 2 minutes. Use of 0.5% Sodium Hypochlorite will be done for flushing the tubing of dental chair waterline and the same solution would be allowed to stay in tubing for 10 minutes followed by water flushing to remove the unwanted biofilm from the tubing surfaces. This procedure would be done at the end of each treatment.

Then operatory will fumigated at the end of all procedures to allow the room to be free of aerosol before it is allowed for use for the subsequent subject. Dental unit would use distilled water in self-contained system, for the study.

i) Primary outcome: microbial colony forming unit Passive sampling will be conducted to assess the index of microbial air contamination as described in other studies (Pasquarella C, et al 2000, Napoli C, et al 2012, Saha R, et al 2017). The method quantifies the microbial flow directly related to the contamination of surfaces coming from microbes that reach critical points by falling on to them. The index of microbial air contamination is based on the count of the microbial fallout on to Petri dishes left open to the air according to the 1/1/1 scheme (for 1h, 1m from the floor, at least 1m away from walls or any obstacle). This index corresponds to the values of CFU calculated from the culture plates of 9 cm diameter. Sealed petri dishes will be transported to where the procedures will be done. Gravity settle plates using tryptic soy agar in 9cm Petri dishes will be used to assess the colony count for passive sampling. The index of microbial air contamination will be assessed at rest (in the early morning before the beginning of dental procedures) and in operational of procedures (during procedures) to determine changes in bacterial count due to dental treatment. Five resting and five in operational samples will be taken from each room. Plates will be incubated overnight at 37°C and colony counts will be documented.

ii) Secondary outcome: patient acceptance Patient will complete a self-administered questionnaire to determine their acceptance over the experience to undergo the scaling procedure.

ELIGIBILITY:
Inclusion Criteria:

* BPE score of 2

Exclusion Criteria:

* BPE score of 1, 3 or 4
* Smoker
* Systemic disease

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Total bacterial count | 30 mins
  The index of microbial air contamination is based on the count of the microbial fallout on to Petri dishes left open to the air according to the 1/1/1 scheme (for 1h, 1m from the floor, at least 1m away from walls or any obstacle). This index corresponds to the values of CFU calculated from the culture plates of 9 cm diameter. The index of microbial air contamination will be assessed at rest (before the beginning of dental procedures) and in operational of procedures (during procedures) to determine changes in bacterial count due to dental treatment.

SECONDARY OUTCOMES:
Patient acceptance of dental procedure | 1 treatment session, which is about 30 mins
  The patient will be given a questionnaire after the treatment to assess their acceptance over the treatment procedure i.e. having scaling procedure by the method (control or interventional). The perception will assessed using Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No